CLINICAL TRIAL: NCT03985163
Title: Capturing Opioid Use Disorder Electronically & Patient Reported Outcomes
Brief Title: Patient Reported Outcomes for Opioid Use Disorder
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Drug Abuse Treatment Clinical Trials Network (Network); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2000024667; 3UG1DA015831-17S1 (NIH)
Record Dates: First submitted 2019-06-10; First posted 2019-06-13 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Opioid-use Disorder; Overdose of Opiate; Patient Participation
Keywords: Patient Reported Outcomes; Clinical Data Research; Electronic Health Records
MeSH Terms: conditions — Opioid-Related Disorders; Opiate Overdose; Patient Participation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patient Reported Outcomes Electronic Survey — This study does not include a drug, test, behavioral or medical procedure intervention; participants will be asked to complete three surveys

SUMMARY:
The goal of the project is to build a clinical data research infrastructure that will begin to enhance capacity to use electronic health record (EHR) data and patient reported outcomes measures (PROs) to conduct opioid related research in emergency departments (EDs). 200 adult patients with a history of non-medical opioid use, opioid use disorder, or acute opioid overdose will be enrolled and will be asked to complete three PRO surveys (baseline, 3 days post ED discharge, and 30 days post discharge).

ELIGIBILITY:
Inclusion Criteria:

* Adult patient presenting to the Yale New Haven Hospital York Street Campus emergency department
* History of opioid use disorder or non-medical use of opioids, as measured by screening assessment OR receiving treatment for opioid overdose
* Willingness and ability to complete electronic surveys via a smartphone or computer

Exclusion Criteria:

* <18 years of age
* Inability to communicate in English
* Inability to provide consent (for example, due to psychosis, intoxication, severe mental illness or other reason)
* Transfer from the ED for psychiatric evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult ED patients with OUD or non-medical opioid use, or those who are being treated for opioid overdose.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2019-06-07 (Actual); Primary Completion 2020-02-16 (Actual); Study Completion 2020-02-16 (Actual)

PRIMARY OUTCOMES:
Willingness to share EHR data with researchers | once: at screening and enrollment
  The proportion of people who qualify for study criteria and enroll in the study
Electronic survey response | once: 3 day follow-up survey
  Response rate to patient reported outcomes via electronic follow-up survey

SECONDARY OUTCOMES:
Treatment Effectiveness Assessment | once: 3 day follow-up survey
  Treatment Effectiveness Assessment (TEA) elicits patient responses that help the patient and the clinician quickly gauge patient progress in treatment and in recovery, according to the patients' sense of what is important within four domains (substance use, health, lifestyle, and community) established by prior research
Treatment Effectiveness Assessment | once: 30 day follow-up survey
  Treatment Effectiveness Assessment (TEA) elicits patient responses that help the patient and the clinician quickly gauge patient progress in treatment and in recovery, according to the patients' sense of what is important within four domains (substance use, health, lifestyle, and community) established by prior research
ED patients prescribed opioid use disorder medication | once: 3 day follow-up survey
  The proportion of participants prescribed opioid use disorder medication as part of routine emergency medical care
ED patients prescribed opioid use disorder medication | once: 30 day follow-up survey
  The proportion of participants prescribed opioid use disorder medication as part of routine emergency medical care
ED patients referred to substance use disorder treatment | once: 3 day follow-up survey
  The proportion of participants referred for substance use disorder treatment as part of routine emergency medical care
Patients enrolling in substance use disorder treatment | once: 30 day follow-up survey
  The proportion of participants referred for substance use disorder treatment who enroll in substance use disorder treatment
Patients filling opioid use disorder prescriptions | once: 3 day follow-up survey
  The proportion of participants prescribed opioid use disorder medication who fill the opioid use disorder prescription
Patients filling opioid use disorder prescriptions | once: 30 day follow-up survey
  The proportion of participants prescribed opioid use disorder medication who fill the opioid use disorder prescription
Lost-to-follow-up | Up to 5 months
  Lost-to-follow-up rates
Electronic survey response | once: 30 day follow-up survey
  Response rate to patient reported outcomes via electronic follow-up survey

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Hawk, MD, Principal Investigator — Yale University School of Medicine Department of Emergency Medicine
Locations (1):
- Yale New Haven Hospital - York Street Campus - Emergency Department, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Hawk K, Malicki C, Kinsman J, D'Onofrio G, Taylor A, Venkatesh A. Feasibility and acceptability of electronic administration of patient reported outcomes using mHealth platform in emergency department patients with non-medical opioid use. Addict Sci Clin Pract. 2021 Nov 10;16(1):66. doi: 10.1186/s13722-021-00276-0. PMID 34758881

DOCUMENTS (1):
  • Informed Consent Form (2019-04-26): https://cdn.clinicaltrials.gov/large-docs/63/NCT03985163/ICF_000.pdf